CLINICAL TRIAL: NCT01423045
Title: Association Between Urine Concentration Ability and the Progression of Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Benaya Rozen-Zvi (Other)
Responsible Party: Sponsor-Investigator, Benaya Rozen-Zvi, attending nephrologist pre dialysis clinic Dan petach-tiqua county, Meir Medical Center
Organization: Meir Medical Center (Other)
Other Study IDs: UCONC
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Urine osmolarity; Glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is that urine concentrating ability can predict the rate of kidney function decline.

Patients with kidney disease at the investigatorsclinic will be asked to give first morning urine sample and osmolarity will be measured. The investigators will follow up kidney function decline and check if there is association with urine osmolarity.

DETAILED DESCRIPTION:
Design:

Prospective observational study

Setting:

Predialysis clinic.

Participants:

We will include adults >18 years providing signed informed consent.

Inclusion:

Patients with CKD and estimated GFR of less then 50 mL per minute estimated by the short MDRD equation base on two creatinine values taken at least two weeks apart and are not getting steroids or immunosuppressive medication as treatment for their primary kidney disease.

Exclusion:

1. Life expectancy of less then 6 month.
2. Expected to start renal replacement therapy within 3 month.
3. Acute or acute on chronic renal failure with reversible component.
4. Treatment with AVP inhibitors.
5. Chronic hyponatremia (Na+<135 in two measurement two weeks apart).
6. Primary polydipsia.
7. Inability to give informed consent.
8. Clinical hypovolemia.

Outcomes:

Primary outcomes:

Rate of GFR decline as assessed by short MDRD equation with at least three measurements at least three month apart.

. Secondary efficacy

1. Rate of ESKD define as need RRT.
2. Overall mortality.
3. ESKD and overall mortality.
4. Blood pressure as assessed by clinic measurement.
5. Protein creatinine ratio in random urine sample.
6. Hemoglobin level.
7. Need for erythropoietin treatment.
8. Blood level of 25OH vitamin D and 1,25OH vitamin D.
9. PTH, calcium and phosphate level.
10. The occurrence of edema by physical evaluation.

Predefined subgroup analysis:

1. Diabetic patients.
2. Patients treated with diuretics.

Sample size:

We will need to recruit about 200 patients.

Statistical methods:

We will use linear regression analysis with 95% CI for the continuous variable. And chi square for dichotomous variable.

Data collection and trial flow:

All patients in predialysis clinic of Dan district of "Kupat holim clalit" will be screen. Patients fulfilling inclusion criteria will be approached by trial investigator for informed consent and trial recruitment. For patients fulfilling inclusion criteria that will not consent to participate we will be record name and ID without further details. Consenting patients will bring the three samples of first voided urine of the morning for osmolarity, PH, sodium, potassium and chloride.

Patient recruitment:

Baseline data collection:

Collection of data will include baseline conditions, primary kidney disease, current medications, clinical evaluation for edema and blood pressure.

Laboratory results will include creatinine, urea, sodium, potassium, GFR assessed by short MDRD equation, protein creatinine ratio in random urine sample Hb level, vitamin D level calcium, phosphorus and PTH.

Follow-up and outcome data collection:

1. Creatinine, estimated GFR, urea, sodium, potassium chloride, hemoglobin and protein creatinine ratio in random urine sample at least every three month
2. Clinical assessment for edema and blood pressure ant least every three month.
3. Time to initiation of dialysis or transplantation.
4. Mortality of any cause and cardiovascular mortality.
5. Hospitalization for any cause and the length of hospital stay.
6. The need for ESA treatment and ESA dose will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD and estimated GFR of less then 50 mL per minute estimated by the short MDRD equation base on two creatinine values taken at least two weeks apart and are not getting steroids or immunosuppressive medication as treatment for their primary kidney disease.

Exclusion Criteria:

1. Life expectancy of less then 6 month.
2. Expected to start renal replacement therapy within 3 month.
3. Acute or acute on chronic renal failure with reversible component.
4. Treatment with AVP inhibitors.
5. Chronic hyponatremia (Na+<135 in two measurement two weeks apart).
6. Primary polydipsia.
7. Inability to give informed consent.
8. Clinical hypovolemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD and estimated GFR of less then 50 mL per minute.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
eGFR slope | 12 month
  Creatinnie value will be measured at least every three month and eGFR will be calculated by MDRD equation. A regression line will be plotted against time and the eGFR slope will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Benaya Rozen-Zvi, MD, Principal Investigator — General health services - Dan Petach tiqua county
Locations (1):
- Pre dialysis clinic Dan Petach Tiqua county General health service, Ganey Tiqua, Israel